CLINICAL TRIAL: NCT02753647
Title: A Prospective, Single Arm, Open-label, Phase II Study of Chidamide in Combination With R-CHOP in the Treatment of de Novo, Elderly, High-risk Diffuse Large B-cell Lymphoma
Brief Title: Chidamide Plus R-CHOP in Elderly DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-CHOP
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide plus R-CHOP (Experimental): Rituximab 375 mg/m2 IV d1 Cyclophosphamide 750mg/m2 IV d2 Doxorubicin 50mg/m2 IV d2 Vincristine 1.4 mg/m2 IV d2 Prednisone 60 mg/m2 PO d2-6 Chidamide 20mg/d PO d1, 4, 8, 11 Frequency every 21 days for 6 cycles
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Chidamide

INTERVENTIONS:
Drug: Rituximab
Drug: Cyclophosphamide
Drug: Doxorubicin
Drug: Vincristine
Drug: Prednisone
Drug: Chidamide

SUMMARY:
This is a prospective, single-arm, open-label phase II study of Chidamide in combination with R-CHOP in the treatment of de novo, elderly, high-risk diffuse large B cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diffuse large B-cell lymphoma, CD20 positive
* Age 61-75 years
* ECOG 0,1,2
* Life expectancy>6 months
* Informed consented
* IPI>1

Exclusion Criteria:

* Chemotherapy before
* Stem cell transplantation before
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary CNS lymphoma
* LVEF≤50%
* Lab at enrollment (Unless caused by lymphoma) Neutrophile<1.5*10^9/L Platelet<75*10^9/L ALT or AST >2*ULN,AKP or bilirubin >1.5*ULN Creatinine>1.5*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Not able to comply to the protocol for mental or other unknown reasons
* Pregnant or lactation
* HIV infection
* If HbsAg positive, should check HBV DNA, DNA positive patients cannot be enrolled. If HBsAg negative but HBcAb positive (whatever HBsAb status), should check HBV DNA,DNA positive patients cannot be enrolled.

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)

SECONDARY OUTCOMES:
Progression free survival rate | 2 year
Overall survival rate | 2 year
Overall response rate | 21 days after 6 cycles of treatment (each cycle is 21 days)
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Each cycle of treatment and then every 3 months for 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang MC, Fang Y, Wang L, Cheng S, Fu D, He Y, Zhao Y, Wang CF, Jiang XF, Song Q, Xu PP, Zhao WL. Clinical efficacy and molecular biomarkers in a phase II study of tucidinostat plus R-CHOP in elderly patients with newly diagnosed diffuse large B-cell lymphoma. Clin Epigenetics. 2020 Oct 23;12(1):160. doi: 10.1186/s13148-020-00948-9. PMID 33097085